CLINICAL TRIAL: NCT03356782
Title: Safety and Efficacy Evaluation of 4th Generation Safety-engineered CAR T Cells Targeting Sarcomas
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17016
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Sarcoma; Osteoid Sarcoma; Ewing Sarcoma
Keywords: CART; PD-1; PDL-1; CTLA-4; sarcoma; solid tumor
MeSH Terms: conditions — Sarcoma; Bone Neoplasms; Sarcoma, Ewing; Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sarcoma-specific CAR-T cells (Experimental): Peripheral blood mononuclear cells (PBMCs) of patients who have CD133, GD2, Muc1, CD117 or other marker positive sarcoma will be obtained through apheresis, and T cells will be activated and modified to sarcoma-specific CAR-T cells.
  Interventions: Biological: Sarcoma-specific CAR-T cells

INTERVENTIONS:
Biological: Sarcoma-specific CAR-T cells — 1 infusion, for 1x10^6~1x10^7 cells/kg via IV

SUMMARY:
The aim of this clinical trial is to assess the feasibility, safety and efficacy of CAR T cells immunotherapy in patients who have sarcoma that is relapsed or late staged. Another goal of the study is to assess the safety and efficacy of the therapy that combines CAR T cells and IgT cells to treat sarcoma.

DETAILED DESCRIPTION:
Patients with late staged and/or recurrent sarcoma have poor prognosis despite complex multimodal therapy. Therefore, novel curative approaches are needed.This study will combine two different ways to fight sarcoma: antibodies and CAR-T cells. Several immune checkpoint antibodies have been examined on various tumors with good outcomes. Sarcoma is known to express increased levels of surface antigens that can be targeted by CAR-T cells. Thus, in this study, the 4SCAR-IgT cells targeting sarcoma surface antigens will be infused in dose escalation cohorts.This study will assess the feasibility, safety, efficacy and side effects of CAR T cells immunotherapy in patients who have sarcoma that is relapsed or late staged.

ELIGIBILITY:
Inclusion Criteria:

1. Stage Ⅲ，Ⅳ sarcoma patients or recurrent sarcoma patients;
2. Age: ≥ 18 and ≤65 years of age at the time of enrollment;
3. At least 4 weeks since any chemotherapy or radiotherapy and at least 1 week since immunosuppressive therapy such as using steroid hormone before enrollment;
4. Side effects of chemotherapy have been well managed;
5. Malignant cells are target antigen positive(higher than ++) confirmed by IHC, quantitative PCR or sequencing;
6. Karnofsky /jansky score of 50% or greater;
7. Expected survival > 6 weeks;
8. ANC≥ 1×10^6/L，PLT ≥ 1×10^8/L;
9. Pulse oximetry of≥90% on room air；
10. Adequate hepatic function,defined as aspartate aminotransferase(AST)< 5 times upper limit of normal(ULN),serum bilirubin < 3 times ULN;
11. Adequate renal function,defined as serum creatinine less than 2 times ULN,if serum creatinine more than 1.5 times ULN,creatinine clearance rate test is needed;
12. Patients must have autologous transduced T cells at levels greater than 15%;
13. Sign an informed consent and assent.

Exclusion Criteria:

1. The disease is progresseing rapidly;
2. The patient is receiving therapy of other new drugs;
3. Evidence of tumor potentially causing airway obstruction;
4. Epilepsy history or other CNS diseases;
5. Patients who need immunosuppressive drugs because of GVAD;
6. History of long QT syndrome or severe heart diseases;
7. Uncontrolled active infection;
8. Active hepatitis B virus,hepatitis C virus and HIV infection;
9. Receiving systemic corticosteroid 2 weeks before enrollment except for inhaled steroids;
10. Previous treatment with any gene therapy;
11. Creatinine>2.5mg/dl or ALT/AST>3 times normal or bilirubin>2.0 mg/dl;
12. Patients who have other uncontrolled diseases would preclude participation as outlined;
13. Pregnant or lactating women;
14. Patients previously experienced toxicity from cyclophosphamide;
15. Patients who have CNS sarcoma;
16. In condition that may bring risks to subjects or interference to clinical trials.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of CART cells in patients using CTCAE version 4.0 standard to evaluate the level of adverse events | 3 months
  Physiological parameter (measuring cytokine response)

SECONDARY OUTCOMES:
Persistence and proliferation of CART cells in patients | 3 months
  The expansion and functional persistence of CART cells in the peripheral blood of patients will be measured by qPCR on Day 7, 14, 21, 28, 60 and 90 after infusion.

OTHER OUTCOMES:
Anti-tumor effects | 1 year
  Objective response, such as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, PhD, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903